CLINICAL TRIAL: NCT02820636
Title: Treatment for Latino/a Adolescents With Suicidal Behavior
Brief Title: Latino/a Adolescents With Suicidal Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Yovanska Duarte-Velez, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH097772 (NIH)
Record Dates: First submitted 2016-03-28; First posted 2016-07-01 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Suicide
Keywords: Suicidal ideation; Suicide attempt; Latinx teens
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- InVita (Experimental): Participants receive the Socio-Cognitive Behavior Therapy (S-CBT) treatment.
  Interventions: Behavioral: S-CBT
- Treatment as Usual (Active Comparator): Intensive outpatient therapy of standard care for adolescents and their parents
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: S-CBT — The SCBT-SB protocol has 3 phases. Phase I, which is fixed (core sessions), includes 9 sessions (1 family, 5 individual & 3 caretakers sessions). Topics include: understanding the suicidal crisis, identity in adolescence, chain analysis, communication skills, the power of thought and decision making, parenting skills, rearing in a different culture, and family communication. Phase II is flexible and consists of coping skills modules (thoughts, emotional regulation, social interactions, activities, substance abuse, family communication & trauma). The treatment plan is adjusted to adolescents' needs. Family and primary caregiver sessions are flexible, depending on the family/caregivers' needs. Participants have received an adequate course of treatment if they at least complete the core sessions. This protocol should take 3-6 months. Once the active phase ends, booster sessions are recommended.
  Arms: InVita
Behavioral: Treatment as Usual — Intensive outpatient therapy with teens and their parents using a variety of eclectic treatments that characterize standard care for adolescents.
  Arms: Treatment as Usual

SUMMARY:
The study is about developing the best aftercare treatment possible for Latino/a adolescents who have been hospitalized in a psychiatric unit due to a suicidal crisis (suicidal thoughts or attempts). The treatment's purpose is to help adolescents and their caregivers develop skills to prevent future suicidal crises. Latino/a adolescents usually report more suicidal behavior than other ethnic groups. The question that the investigators want to answer is if a new treatment (socio-cognitive behavioral therapy-(SCBT)) developed to their specific needs, taking into account their culture and aspects of adolescence, performs better than the treatment that they usually receive. Forty six adolescents were recruited from the Bradley Hospital adolescent inpatient unit or the Hasbro Inpatient Medical & Psychiatric Program, or referred to Gateway Healthcare after discharge from other inpatient units in Rhode Island; half of them were assigned randomly to the treatment they would usually receive (TAU) and the other half to the new treatment (SCBT). In both groups, caregivers and adolescents completed questionnaires and interviews before the beginning of treatment and at 3, 6, and 12 months after the treatment begin. Questions to the participants were related to their presenting symptoms, family, social group, problems, and other similar topics. Also, participants were asked about their satisfaction with the treatment they were receiving. The purpose of the questionnaires and interviews are to follow their progress in therapy. At the end, comparisons will be made between the group who participated in TAU and the group who participated in the SCBT, based on the assessment results from the adolescents and caregivers.

DETAILED DESCRIPTION:
The primary aim of the proposed research is to evaluate the feasibility of a socio-cognitive-behavioral therapy protocol for suicidal behavior (SCBT-SB) with Latino/a adolescents in comparison to treatment as usual (TAU). The SCBT-SB protocol was develop in Puerto Rico, but was expand to Latinx populations in U.S. based on a previous qualitative study. The SCBT-SB include developmental and cultural factors in order to optimize treatment outcomes in suicidal Latino/a adolescents. Study design: A pilot randomized controlled trial (RCT) of the SCBT-SB versus TAU was conducted in a real world scenario. Participants were 46 Latino/a adolescents (13-17) admitted to a Psychiatric Unit for suicide ideation or suicide attempts, who were referred to outpatient care, and at least one legal guardian. RCT's primary question is: Is the SCBT-SB protocol feasible in terms of satisfaction, acceptability, recruitment, retention, and therapist adherence? RCT's secondary question is: What is the magnitude of difference in suicidality and psychopathology symptoms between the SCBT-SB and the TAU at three, six, and 12 months following baseline?

ELIGIBILITY:
Inclusion Criteria:

* Latino/a
* Admitted to the inpatient unit for suicidal ideation or suicidal behaviors

Exclusion Criteria:

* Severe psychosis or psychoses independent of depression
* Department of Children and Families (DCYF) involvement
* Status as a ward of the state

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of Suicide Behaviors (attempts, aborted & interrupted attempts, preparatory acts) and Suicide Events (hospitalizations, ER visits) | Change from Baseline to 6 Month (6M) and 12 Month (12M)
  Number of behaviors or events measured using the Columbia Suicide Severity Rating Scale (C-SSRS)
Suicidality | Change from Baseline to 6 Month (6M) and 12 Month (12M)
  Measured using the Suicidal Ideation Questionnaire (SIQ-JR)

SECONDARY OUTCOMES:
Psychiatric Symptoms [Axis I Diagnoses] | Change from Baseline to 6M and 12M
  Axis I diagnoses as evaluated from the Children's Inventory for Psychiatric Syndromes (ChIPS) and Youth Self-Report (YSR)
Depressive Symptoms | Change from Baseline to 6M and 12M
  Level of depressive symptomatology measured using the Children's Depression Inventory (CDI)

CONTACTS AND LOCATIONS:
Overall Officials: 02915 02915, Ph.D., Principal Investigator — Brown University
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States